CLINICAL TRIAL: NCT03765970
Title: Transcultural Validation of MSTS and TESS Questionnaire
Acronym: MSTS-TESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC17_0487
Record Dates: First submitted 2018-06-19; First posted 2018-12-05 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-06

CONDITIONS: Cancer
Keywords: Tumor resection; MSTS; TESS; Soft tissue and bone; Questionnaires
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reference treatment for soft tissue or bone sarcoma is the Monobloc resection surgery, with a margin of one to many millimeters removing the entire tumor leaving no cancer cells, associated or not with other treatments. Other musculoskeletal malignant tumors, some of them with secondary origins (metastases), are treated the same way. Patients with soft tissue and bone tumor could have heavy sequels of this surgery procedure, depending on the localization and size of the initial tumor. Those functional sequels are evaluated by specific questionnaires: the questionnaire TESS for upper limbs and TESS for lower limbs which are completed by the patient (depending on the localization of the tumor) and the questionnaire MSTS which is completed by the medical doctor.

Those English validated questionnaires are frequently used by French surgeons in standard practice as well as scientific research. The translations done have never been validated by an official methodology.

The aim of this trial is to validate the TESS and MSTS questionnaires linguistically, culturally (questions must be adapted for each target population: occidental adults and adolescents population, male and female population and adapted to the current era), and scientifically (repeatability).

The validation of those questionnaires will permit to have functional and reference questionnaires in French language which could be used for the follow up of operated patient in the context of the care and clinical research.

DETAILED DESCRIPTION:
The methodology will follow the guidelines of Dorcas E. Beaton, Claire Bombardier, Francis Guillemin and Marcos Bosi Ferraz (approved in particular by the American Academy of Orthopedic Surgeons):

Step 1: Author's agreement Step 2: Translation with cultural adaptation in addition to literal translation Step 3: 2 first translations English to French (2 different translators T1 and T2) Step 4: Synthesis (T12) Step 5: 2 reverse translations of T12 French to English (BT1 and BT2) Step 6: Submission to a committee of experts of the final translation Step 7: Clinical study based on a sample of patients (questionnaires, interview and analysis of the distribution of responses) The investigators planned the recruitment of 250 adults and adolescents patients over 15 years old, who will answers to the questionnaires (MSTS-TESS) as well as control-questionnaires (WOMAC or DASH) during a follow-up consultation, in Nantes, Rennes, Tours or Marseille centers. A study of repeatability will be performed with 30 to 50 patients for whom 2 filling will be necessary, the first time during the consultation and the second time at home, 15 days later.

ELIGIBILITY:
Inclusion Criteria:

* Major Patients who has accepted and be informed of the protocol or minor patient over 15 years old who has accepted and be informed of the protocol, with the agreement of one legal representative
* Patients over 15 years old who had a surgical procedure for a musculoskeletal tumor which could result in functional sequels. (at the appreciation of the surgeon)
* Patients in the capacity to answer and understand the questionnaire and for whom the French is the native language

Exclusion Criteria:

* Patients refusing to participate
* Patient under guardianship
* Patient inappropriate for entry into this study according to the judgment of the investigator

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population is adults and adolescents aged 15 and over operated on tumor surgery that can lead to functional sequelae.
  These patients will be evaluated at the post-surgical consultation or during a consultation of followed regardless of the seniority of the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Validation of psychometric properties of questionnaire MSTS in French translation | one day

SECONDARY OUTCOMES:
Define questionnaires content validity : evaluation of translation quality (expert consensus). | one day
  After the 2 translations and retrotranslations of the questionnaires adapted to the present time and the target population, an expert committee composed of health professionals meets with the aim of proposing a unified version. This latest version is subject to the approval of the original authors.
Define face validity : evaluate the comprehension of the questionnaire by 5 to 10 patients (qualitative analysis) | one day
Define questionnaires construction validity: coherent evolution of scoring with the clinical status of the patients (ANOVA) | 3 months (after study completion)
Define criteria validity: coherence with other scores (correlation with WOMAC-long form >0.4) | one day
Define score reliability: intern coherence and responses coherence (Cronbach's alpha > 0.7 and Loevinger's H > 0.3) | 3 months (after study completion)
Verify the repeatability of the questionnaire MSTS on 30 to 50 patients : concordance between answers of two surgeons on the same consultation | one day
Define criteria validity for upper limbs: coherence with DASH score (correlation with DASH >0.4) | one day
Verify the repeatability of the questionnaire TESS on 30 to 50 patients: concordance between answers of the same patient completing twice the same questionnaires (first during the consultation and then 15 days after at home). | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin BRULEFERT, Dr, Principal Investigator — Nantes University Hospital
Locations (5):
- France (5):
  - Marseille University Hospital, Marseille
  - Nantes University hospital, Nantes
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours